CLINICAL TRIAL: NCT02143999
Title: An Observational Study of BRAF Inhibitors Effectiveness in Patients With Newly Diagnosed Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29031
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the effectiveness of BRAF inhibitors and current therapies in patients with newly diagnosed metastatic melanoma with or without BRAF V600 mutation. Patients will be treated per the locally approved therapeutic options in clinical practice. The observation period for each patient will be up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age at diagnosis
* Histologically confirmed new diagnosis of unresectable or metastatic melanoma
* Patients with tumor samples available for assessment of BRAF V600 mutation

Exclusion Criteria:

* Prior systemic therapy for metastatic disease
* Participation in interventional clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed unresectable or metastatic melanoma
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Best Overall Response Rate (BORR) | 2 years
Time to response | 2 years
Duration of response | 2 years
ECOG performance status | 2 years
Safety: Incidence of adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Italy (24):
  - Policlinico Ospedaliero Ss Annunziata; U.O. Di Clinica Oncologica, Chieti, Abruzzo
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari, Apulia
  - IRCCS IST. Tumori Fondaz. Pascale; S.C. Oncologia Medica,Melanoma,Immunoterapia E Terapie Innovative, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST);U.O. di Immunoterapia, Meldola, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - Az. Osp. Spedali Civili; Divisione Di Oncologia - Iii Medicina, Brescia, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (Ieo); Unita' Di Ricerca Traslazionale Del Melanoma, Milan, Lombardy
  - Fondazione Del Piemonte Per L'oncologia IRCC Di Candiolo, Candiolo, Piedmont
  - Azienda Sanitaria Ospedaliera s. Croce e Carle; Oncologia Medica, Cuneo, Piedmont
  - Ospedale Maggiore Della Carita; Oncologia Medica, Novara, Piedmont
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Policlinico P. Giaccone; Istituto Di Oncologia, Clinica Medica 1, Palermo, Sicily
  - Ospedale S. Vincenzo; Oncologia Medica, Taormina, Sicily
  - Azienda Sanitaria di Firenze Presidio Palagi - SC Dermatologia II e Fisioterapia Dermatologica, Florence, Tuscany
  - Azlenda Ospendaliero-Universitaria Pisana; C.O. Oncologia 2, Pisa, Tuscany
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
  - Azienda Ospedaliero Universitaria di Ferrara - U.O. Di Oncologia, Cona (FE), Veneto
  - Azienda Ospedaliera di Verona-Policlinico G.B. Rossi; Oncologia Medica, Verona, Veneto